CLINICAL TRIAL: NCT01017107
Title: APCAP - Activated Protein C in Severe Acute Pancreatitis: A Double-blind Randomized Human Pilot Trial
Brief Title: Activated Protein C in Severe Acute Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Kemppainen Esko / M.D. PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HUS 210284
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2009-11

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; treatment; organ failure; activated protein c
MeSH Terms: conditions — Pancreatitis | interventions — Protein C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activated protein C (Experimental)
  Interventions: Drug: Activated protein C

INTERVENTIONS:
Drug: Activated protein C — 24 micrograms/kg/hour intravenously for 96 hours

SUMMARY:
Activated protein C (APC)has been shown to reduce mortality in severe sepsis(Bernard et al. 2001b). The clinical picture of severe acute pancreatitis (AP) is similar to that of sepsis. The investigators conducted a randomised double-blinded placebo-controlled pilot study in AP patients (16+16) with the same dose of APC that has been proven to be efficacious and safe in septic patients.

The aim of the study is to investigate whether the APC replacement therapy diminishes the occurrence and severity of organ dysfunction in patients with severe AP. The effect of APC on inflammatory and hemostatic parameters is also assessed.

DETAILED DESCRIPTION:
The study started in 2003 and was finished in 2007. The study was registered in The Helsinki University Central Hospital study register in 2003.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital within 72 h of the onset of pain.
* Plasma amylase concentration more than three times the upper limit of the normal range and/or CT findings compatible with AP.
* Organ failure and <48h of the onset of the first organ failure

Exclusion Criteria:

* HIV / B- or C hepatitis infection
* Pregnancy or breast feeding
* Active bleeding
* Increased risk of bleeding (thrombocytes <30x10E9/L or INR>3.0
* Gastrointestinal bleeding within 6 weeks or intracranial stroke within 3 months before the study
* Intravenous contrast extravasation or other signs (fresh hematoma) suggesting active hemorrhage within the pancreas or in the peripancreatic area on admission CT scan
* Use of antithrombin III within 12 h
* Use of acetylsalicylic acid or glycoprotein IIB/IA antagonist within 7 days / Thrombolytic therapy within 3 days
* Surgery requiring general or spinal anaesthesia within 12 h
* Previous pancreatic surgery
* Application of an epidural catheter within 48 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint was the number of bleedings, and the primary efficacy endpoint was the change in SOFA between the start of the drug (day 0) and day 5. | 0-60 days

SECONDARY OUTCOMES:
Organ failure free days alive | 0-60 days

CONTACTS AND LOCATIONS:
Overall Officials: Ville Pettilä, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Bernard GR, Vincent JL, Laterre PF, LaRosa SP, Dhainaut JF, Lopez-Rodriguez A, Steingrub JS, Garber GE, Helterbrand JD, Ely EW, Fisher CJ Jr; Recombinant human protein C Worldwide Evaluation in Severe Sepsis (PROWESS) study group. Efficacy and safety of recombinant human activated protein C for severe sepsis. N Engl J Med. 2001 Mar 8;344(10):699-709. doi: 10.1056/NEJM200103083441001. PMID 11236773
- [Derived] Pettila V, Kyhala L, Kylanpaa ML, Leppaniemi A, Tallgren M, Markkola A, Puolakkainen P, Repo H, Kemppainen E. APCAP--activated protein C in acute pancreatitis: a double-blind randomized human pilot trial. Crit Care. 2010;14(4):R139. doi: 10.1186/cc9203. Epub 2010 Jul 27. PMID 20663207